CLINICAL TRIAL: NCT05292430
Title: B2RAD Translational Medicine Study
Acronym: B2RAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohail Rao (Other)
Responsible Party: Sponsor-Investigator, Sohail Rao, President and CEO, DHR Health Institute for Research and Development
Organization: DHR Health Institute for Research and Development (Other)
Other Study IDs: 1551551
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Specimens Are to be Collected From Subjects Who Are Having or Have Had a Fluid or Tissue Removed, a Biopsy or a Blood or Bone Marrow Draw
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — fluid or tissue removed, a biopsy or a blood or bone marrow draw. The specimen requirements are approximately 80 mgs to 1 gm or more of fresh, frozen, or formalin fixed paraffin embedded ("FFPE") viable diseased tissue and up to 700 gms of viable normal tissue (when available). In addition, blood and/or bone marrow specimens may be obtained at diagnosis, during therapy, during remission, or at the time of relapse. Blood collection may range from 2-15tubes or approximately 20 to 150 mLs. Depending on the protocol it may be necessary to collect other biospecimens such as urine, stool, saliva, bronchial lavage, nasal fluids, or fine needle aspirates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biobank: Specimens are to be collected from subjects who are having or have had a surgical or medical procedure (such as fluid or tissue removed, a biopsy or a blood or bone marrow draw). Any subject in which the primary diagnosis of disease was made within the DHR Health System and Any subject choosing to give consent for participation will be included.
  Interventions: Other: Specimen Collection

INTERVENTIONS:
Other: Specimen Collection — collection of diseased and non-diseased tissue, blood, and other body fluids

SUMMARY:
Recent advances in understanding the molecular and cellular pathology of many diseases have resulted in direct benefit to today's patients. The translational research studies that have led to these advances relied on an integrated model of clinical and non-clinical laboratory investigations based on the analysis of human biospecimens that lead directly to drug discovery, drug validation, novel detection assays, and prognostic marker discovery. Translational research provides a unique mechanism to address questions specific to particular tumor or other disease types, biological modifiers and/or mechanisms of action that are essential for the advancement of healthcare. Specimens are to be collected from subjects who are having or have had a surgical or medical procedure (such as fluid or tissue removed, a biopsy or a blood or bone marrow draw). Any subject in which the primary diagnosis of disease was made within the DHR Health System and Any subject choosing to give consent for participation will be included

ELIGIBILITY:
Inclusion Criteria:

1. Any subject choosing to give consent for participation will be included.
2. Any subject in which the primary diagnosis of cancer was made at the DHR Health System.

Exclusion Criteria:

1. Any subject deemed unable to provide legally effective consent.
2. Any pediatric subject where the subject does not freely give his or her assent or where his or her parent/guardian does not give consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Specimens are to be collected from subjects who are having or have had a surgical or medical procedure (such as fluid or tissue removed, a biopsy or a blood or bone marrow draw). Any subject in which the primary diagnosis of disease was made within the DHR Health System and Any subject choosing to give consent for participation will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Collection of diseased and non-diseased tissue, blood, and other body fluids | once
  Collection of diseased and non-diseased tissue, blood, and other body fluids to establish a biobank to evaluate all potential clinically relevant alterations in the diseased cells, cellular components and disease biomarkers. The methods used to identify these alterations include: 1) Creation of novel disease and normal cell lines; 2) Molecular analysis; 3) Protein analysis; and 4) other cellular analyses. These methods may be employed immediately after obtaining the biologic material or at a future date after samples have been stored in a bank.

CONTACTS AND LOCATIONS:
Overall Officials: Sohail Rao, MD, Principal Investigator — DHR Heath Institute for Research and Development
Locations (2):
- United States (2):
  - DHR Health Institute for Research and Development, Edinburg, Texas
  - DHR Health, Edinburg, Texas

IPD SHARING:
Plan to Share IPD: No